CLINICAL TRIAL: NCT03886285
Title: Establish a Scale of Assessment of the Quality of Primary Care in Multi-functional Health Centers and Homes Integrating the Point of View of Complex Patients and Their Caregivers
Brief Title: A Quality Rating Scale for Patients in Complex Situations
Acronym: Qualsoprim_2
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0019
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2021-06

CONDITIONS: Patients in Complex Situations
Keywords: Multimorbidity; Exercise coordinated groups (GECO); Caregivers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Completion of the questionnaire by the patient after consultation with the general practitioner

SUMMARY:
The prevalence of multimorbid patients and complex care is increasing in France and elsewhere in the world. It concerns 60% of the over 65 years old. Comprehensive care, the involvement of the patient and his caregivers appear as the solutions for the management of these new care situations. The structures of multi-professional grouping, developing a coordinated exercise (GECO), appear as the privileged place to take care of these patients. These structures become the main place of exercise in France (improved working conditions for professionals, financial incentives, public policy, etc.); they have shown their ability to formulate patient care protocols, to produce coordinated exercise, to better involve the patient and caregivers in their care. The question of improving the quality of care arises. To date, there is no data on the subject apart from some evaluations mainly medico-economic.

The patient's place in the evaluation showed his interest with the existence of a proven correlation between patient satisfaction in particular and his compliance and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed in the primary care center, able to participate, speaking and understanding French, and being in a complex care situation, benefiting from a multi-professional care (at least two professionals different from the center including the general practitioner).

Exclusion Criteria:

* Patient not in a complex care situation
* Patient followed only by the general practitioner of GECO
* Refusal of participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed in the primary care center and being in a complex care situation, benefiting from a multi-professional care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Construction of the questionnaire. | 1 day
  The main objective of this phase of the protocol is to structure the questionnaire in order to achieve a scale of assessment of the quality of primary care provided within the coordinated exercise groups from the point of view of complex care patients, their caregivers and patients and health professionals. This questionnaire doesn't exist so it has no name.This questionnaire is qualitative and not quantitative, so nos score is expected.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Maison de santé d'Audierne, Audierne
  - Maison de santé de CAVAN, Cavan
  - Maison de santé de Gourin, Gourin
  - Pôle de santé de Lanmeur, Lanmeur
  - Maison de santé du Faou, Le Faou
  - Maison de santé du Vieux Marché, Le Vieux-Marché
  - Maison de santé de LOUARGAT, Louargat
  - Maison de santé de Milizac, Milizac
  - Maison de santé de Moëlan sur Mer, Moëlan-sur-Mer
  - Maison de santé de Pleyben, Pleyben
  - Maison de santé de Plouneour Trez, Plounéour-Trez
  - Maison de santé de Trébeurden, Trébeurden

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.